CLINICAL TRIAL: NCT06883656
Title: The Pharmacokinetics Study of Fotagliptin in Patients with Different Degrees of Renal Insufficiency and Matched Healthy Volunteers with Normal Renal Function
Brief Title: The Pharmacokinetics Study of Fotagliptin in Patients with Different Degrees of Renal Insufficiency
Acronym: RI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL067-C-011; CTR20212745 (Other: NMPA)
Record Dates: First submitted 2025-03-03; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Renal Insuficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- healthy subject (Active Comparator): Matched healthy subjects
  Interventions: Drug: SAL067
- Mild renal insufficiency (Experimental): Mild renal insufficiency was GFR by 60 to 89 mL/min.
  Interventions: Drug: SAL067
- Moderate renal insufficiency (Experimental): Moderate renal insufficiency was GFR by 30 to 59 mL/min.
  Interventions: Drug: SAL067

INTERVENTIONS:
Drug: SAL067 — Fasting oral test drug 12mg

SUMMARY:
The trial was designed in a single dose, open, non-randomized, multi-dose parallel control group. The study of patients were mild and moderate renal insufficiency, and matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 (including 18 and 75 years old), both male and female;
2. Weight: male ≥ 50 kg, female ≥ 45 kg; BMI in the range of 18 to 30 kg/m2 (including 18 and 30 kg/m2);
3. During screening, the glomerular filtration rate (GFR) met the staging criteria of renal insufficiency or normal renal function in the corresponding group;
4. The subjects can communicate well with the researchers, fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign a written informed consent.
5. During screening, the investigators judged that the kidney disease of the subjects was stable from 4 weeks before screening to the end of the study, and GFR did not change significantly;
6. Patients who had not taken or were on stable medication for renal insufficiency and/or other comorbiditions during the 4 weeks prior to screening and agreed to continue treatment during the study period;
7. Patients with diabetes who have not used hypoglycemic drugs in the 4 weeks prior to screening, or who are receiving stable antidiabetic therapy (including lifestyle interventions, use of stable doses of drugs, except for prohibited drugs described in the trial protocol) and agree to continue treatment during the study period.

Exclusion Criteria:

1. People who are known to be allergic to DPP-4 inhibitors or drug excipients in this study;
2. Previous medication history:

   1. Use of DPP-4 enzyme inhibitors or similar within 2 weeks prior to screening;
   2. Inhibitors or inducers of the CYP 2D6 enzyme used within 30 days prior to screening or required during the trial;
3. Vaccination within 4 weeks prior to screening;
4. Pregnant or lactating women; The subject and his or her spouse or partner have plans to become pregnant, or plan to donate sperm or eggs, or do not agree to an acceptable and effective method of contraception within 3 months of dosing;
5. Hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, HIV antigen antibody composite test any item is positive。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics | 8 day
  Peak blood concentration (Cmax)
Pharmacokinetic characteristics | 8 day
  Area under the curve from 0 to the last time point t (AUC0-last)
Pharmacokinetic characteristics | 8 day
  Area under the curve from 0 to infinity (AUC0-inf)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Hu C, Cao X, Men Y, Wang Y, Zhang R, Guan H, Shi L, Liu F, Miao J. Pharmacokinetics, Pharmacodynamics and Safety of Fultagliptin Benzoate Tablets, a DPP-4 Inhibitor, in Patients With Varying Degrees of Renal Insufficiency and Matched Healthy Volunteers: A Phase I Clinical Trial. Clin Pharmacokinet. 2026 Feb 9. doi: 10.1007/s40262-026-01622-8. Online ahead of print. PMID 41661440